CLINICAL TRIAL: NCT01906177
Title: A Prospective Munti-center Study on VANGUARD™ PS Total Knee Replacement System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: INT.CR.GK5
Record Dates: First submitted 2013-01-07; First posted 2013-07-24 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis; Posttraumatic Deformity
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of this pilot clinical study include:

* Evaluate clinical outcomes and quality of life on patients who received Vanguard PS Total Knee in Korean population
* Evaluate safety of Vanguard PS Total Knee in Korean population

DETAILED DESCRIPTION:
This study is a prospective, single cohort, multi-center study of Vanguard PS system and will be conducted in Korea with 2 institutions. The study will be conducted over a period of 10 years. Patients will be followed at immediate post-op, 6 weeks, 6 months and 1 year, 3 years.

Total of 2 sites will be involved in this study. 50 cases on each sites and total of 100 subjects will be enrolled in the study.

Primary end-point will be KSS at 1 year post op and secondary end-points are Survivorship of the product, KSS, EQ5D, High-Flexion Knee Score, Radiographic Assessment, and any kind of complication including lost to follow up.

ELIGIBILITY:
Inclusion Criteria:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis, where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure
* Need to obtain pain relief and improve function
* Ability and willingness of the patient to follow instructions, including control of weight and activity level
* A good nutritional state of the patient, and
* The patient must have reached full skeletal maturity (at least 18 years old).

Exclusion Criteria:

* infection
* sepsis
* osteomyelitis
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total 100 cases
  each site of 6 sites delegated to enroll 50 cases each
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
American Knee Society Score | 1 year Post Op
  Primary Endpoint: Knee Society Score (KSS) at 1 Year Postop

SECONDARY OUTCOMES:
Survivorship | 3 years post op
  To access the number of patients with implants
EQ-5D | 3 year post op
  Quality of life on patients
Radiographic Assessment | 3 year Post Op
  Access on subsidence, migration, and radiolucency
Complications | 3 year Post Op
  Any AEs to patients

CONTACTS AND LOCATIONS:
Overall Officials: Young Joon Choi, PHD, Principal Investigator — Gangneung Asan Hospital; Jong Keun Seon, PHD, Principal Investigator — Chonnam National University Hospital
Locations (2):
- South Korea (2):
  - Gangneung Asan Hospital, Gangneung-Si, Gangwon-do
  - Chonnam National University Hwasun Hospital, Jeongnam, Jeollanam-do

IPD SHARING:
Plan to Share IPD: No